CLINICAL TRIAL: NCT00197223
Title: A Randomized, Double-blind, Placebo-controlled, Post-marketing Phase III Study to Evaluate the Efficacy of GSK Biologicals' Influenza Vaccine (Fluarix™) Administered Intramuscularly in Adults.
Brief Title: Post-marketing Study to Evaluate the Efficacy of Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 104438
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: Influenza vaccine

SUMMARY:
As a result of the recent supply shortages in the U.S., as well as an anticipated increase in demand during the coming years, GSK Biologicals is pursuing licensure of Fluarix in the U.S. under the accelerated approval process; marketing approval most likely will be granted before the start of this clinical trial. GSK proposes to support U.S. licensure of Fluarix with this confirmatory post-marketing study. The purpose of the study is to evaluate the efficacy of a single dose of Fluarix in preventing influenza in adults during the 2005/2006 Influenza season.

ELIGIBILITY:
Inclusion Criteria:

* A male or female age between, and including, 18 and 64 years of age at the time of the vaccination.
* Written informed consent obtained from the subject.
* Availability to follow up by phone during the study period.
* Female subjects must be of non-childbearing potential, i.e. either surgically sterilized or one year post-menopausal. If subject is of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination. She must also have a negative pregnancy test at study entry and must agree to continue such precautions for two months after vaccination.

Exclusion Criteria:

* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine including egg, chicken protein, formaldehyde, thimerosal, gentamicin sulfate or sodium deoxycholate.
* Acute disease at the time of enrollment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature < 37.5°C).
* Pregnancy
* Chronic disorders of the pulmonary or cardiovascular system, including asthma
* History of requiring regular medical follow-up or hospitalization during the preceding year because of chronic metabolic diseases (including diabetes mellitus), renal dysfunction, hemoglobinopathies, or immunosuppression (including immunosuppression caused by medications or by human immunodeficiency virus.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6213 (Actual)
Dates: Start 2005-09; Primary Completion 2005-10 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Incidence of culture confirmed influenza A and/or B during the surveillance period

SECONDARY OUTCOMES:
Efficacy: Incidence of ILI, Number of days of fever, days of school/work absenteeism, hospitalization related to influenza illness, Incidence of pneumonia, Incidence of PCR confirmed influenza A and/or B

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Beran J, Wertzova V, Honegr K, Kaliskova E, Havlickova M, Havlik J, Jirincova H, Van Belle P, Jain V, Innis B, Devaster JM. Challenge of conducting a placebo-controlled randomized efficacy study for influenza vaccine in a season with low attack rate and a mismatched vaccine B strain: a concrete example. BMC Infect Dis. 2009 Jan 17;9:2. doi: 10.1186/1471-2334-9-2. PMID 19149900
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104438 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register